CLINICAL TRIAL: NCT06319404
Title: A Multiomics-based Study of the Immune Function of Colorectal Cancer Lymph Nodes
Brief Title: Immune Function of Colorectal Cancer Lymph Nodes
Status: Not yet recruiting | Type: Observational
Sponsor: Shanxi Province Cancer Hospital (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2022YFC2505700
Record Dates: First submitted 2024-01-19; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer; Lymph Node
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- negative lymph node
- postive lymph node

INTERVENTIONS:
Other:

SUMMARY:
Lymph nodes are very important immune organs in the human body and play an important role in the physiological and pathological activities of the body, especially in anti-tumor immunity. The role of regional draining lymph nodes in the development of colorectal cancer is still unknown. In this study, the role of lymph nodes in the development of colorectal cancer was investigated through multicenter and multi-omics data.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III colorectal cancer patients undergoing radical surgery
* Complete imaging, pathology and genetics multi-omics data available
* 18-75 years old

Exclusion Criteria:

* Patients with preoperative neoadjuvant therapy
* Patients with incomplete clinical information
* Patients with other malignant tumors
* Patients with acute infections or untreated chronic infections

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stage I-III colorectal cancer patients undergoing radical surgery with complete clinical imaging, pathology, and genetic data.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the difference of immune pathway activation in tumor-draining lymph node based on genomics | 2024.04-2026.04
  BULK-RNA sequencing was performed on tumor draining lymph nodes to detect the activation of immune pathways in lymph nodes and explore the differences between them
To investigate the relationship between the type and number of immune cells in tumor draining lymph nodes and the activation of immune pathways is based on pathomics | 2024.04-2026.04
  Multiple immunohistochemistry was used to identify the type and number of immune cells and to explore the relationship between the activation state of immune pathways
The immune function of tumor draining lymph nodes of colorectal cancer patients was previously identified based on radiomics | 2024.04-2026.04
  Preoperative imaging data (CT, MRI) of patients were collected, and information in the images was extracted based on artificial intelligence algorithms. Predictive models were constructed to identify patients with good or bad immune function before surgery and guide subsequent treatment

IPD SHARING:
Plan to Share IPD: No